CLINICAL TRIAL: NCT00583921
Title: Randomized Study of Ventricular Rate Regularization for Improved Quality of Life in Patients With Congestive Heart Failure and Atrial Fibrillation.
Brief Title: Ventricular Rate Regularization for Improved Quality of Life in Patients With CHF and AF
Acronym: VRR
Status: Withdrawn | Type: Observational
Why Stopped: no subjects enrolled
Sponsor: University of California, Davis (Other)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 200614770
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Congestive Heart Failure; Atrial Fibrillation
Keywords: Atrial Fibrillation; ICD; BiV ICD; CHF; Congestive Heart Failure; AF
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Single center investigator initiated sponsored by Guidant Boston Scientific Corp. to evaluate the benefit of ventricular rate regularization (VRR) in patients with congestive heart failure (CHF) and significant atrial fibrillation (AF) burden.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-85 years old
* Be willing and able to give informed consent
* Patient currently has a CRT-D or ICD with > 20% atrial fibrillation burden as recorded by defibrillator follow up report or a history of atrial fibrillation prior to implant.
* Patient has the ability to complete a Six minute walk test with the only limiting factors to be fatigue or shortness of breath.

Exclusion Criteria:

* Expected mortality less than 6 months due to non-cardiac causes.
* Pregnant women.
* Creatinine greater than or equal to 2.5 mg/dl.
* Anemia (HCT less than 30)
* COPD causing significant dyspnea
* Orthopedic problems affecting 6 minute walk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a new Guidant ICD/ CRT-D: Indication for CRT-D and ICD with history of atrial fibrillation. Patients with new implants will not be enrolled until their three month follow up visit in the pacemaker clinic.
  Patients currenlty implanted with a Guidant ICD/ CRT-D: More than 20% atrial fibrillation burden as recorded by defibrillator follow up report or with history of atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Improved quality of life, reduced emergency room visits and hospitalization for congestive heart failure symptoms. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srivatsa, MD, Principal Investigator — U C Davis Medical Center